CLINICAL TRIAL: NCT06750341
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Different Doses of QLC7401 in Patients With Primary Hypercholesterolemia or Mixed Hyperlipidemia With Poorly Controlled Low-density Lipoprotein Cholesterol (LDL-C) Elevated on Optimized Lipid-lowering Therapy
Brief Title: Study of QLC7401 in the Treatment of Primary Hypercholesterolemia or Mixed Hyperlipidemia With Elevated LDL Cholesterol
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLC7401-201
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Primary Hypercholesterolemia or Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QLC7401 100mg (Experimental): QLC7401 100 mg subcutaneous injection
  Interventions: Drug: QLC7401
- QLC7401 300mg (Experimental): QLC7401 300 mg subcutaneous injection
  Interventions: Drug: QLC7401
- QLC7401 500mg (Experimental): QLC7401 500 mg subcutaneous injection
  Interventions: Drug: QLC7401
- Placebo (Placebo Comparator): Placebo 100/300/500 mg subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QLC7401 — QLC7401 combined with lipid-lowering agents
  Arms: QLC7401 100mg; QLC7401 300mg; QLC7401 500mg
Drug: Placebo — Placebo combined with lipid-lowering agents
  Arms: Placebo

SUMMARY:
To evaluate the efficacy, safety, pharmacodynamics and immunogenicity of QLC7401 subcutaneous administration in patients with primary hypercholesterolemia or mixed hyperlipidemia with poorly controlled LDL-C elevated on optimized lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years of age.
* Serum LDL-C ≥1.8mmol/L for ASCVD participants or ≥2.6mmol/L for other participants at screening.
* Fasting TG <400mg/dL (<4.5mmol/L) at screening.
* Stable lipid-lowering therapy for ≥4 weeks at randomization.
* Understand the study procedures and methods, volunteer to participate in the study, and sign the informed consent.

Exclusion Criteria:

* Having the following diseases or treatment history: (1) cardiac function as defined by the New York Heart Association (NYHA) grade II-IV at screening or randomization or latest detected LVEF<30%; (2) CVD events within 3 months; (3) uncontrolled severe hypertension; (4) previous diagnosis of familial hypercholesterolemia; (5) have known allergic reaction to experimental drug, or have severe allergic reaction to other drugs; (6) inadequate organ functions or malignancy history; (7) prior exposure to other RNA inhibitors within 2 years.
* Any of the laboratory indicators met the following criteria at screening or at randomization: (1) ALT or AST exceeding 2 times the upper limit of normal (ULN), or total bilirubin exceeding 1.5 times ULN; (2) creatine kinase (CK) exceeding 3 times ULN; (3) TSH is less than the lower limit or normal (LLN) or exceeds 1.5 times ULN.
* General conditions: (1) male or female participants who do not agree to use high-efficiency contraceptives during the trial and for 6 months after the last dosing; (2) women who are pregnant or lactating.
* The investigator determines that the participants have poor compliance or have any factors that may prevent them from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage changes in LDL-C from baseline to Day 180 and Day 270 | 80 days and 270 days

SECONDARY OUTCOMES:
Percentage changes in LDL-C from baseline at each subsequent visit to Day 360 | 360 days
Value changes in LDL-C from baseline at each subsequent visit to Day 360 | 360 days
Percentage changes in PCSK9 from baseline at each subsequent visit to Day 360 | 360 days
Value changes in PCSK9 from baseline at each subsequent visit to Day 360 | 360 days
Percentage changes in non-HDL-C, Apo B, TC/HDL-C, Apo A1, Apo B/Apo A1, Lp (a), and TG from baseline to Day 180, Day 270, and Day 360 | 360 days
Value changes in non-HDL-C, Apo B, TC/HDL-C, Apo A1, Apo B/Apo A1, Lp (a), and TG from baseline to Day 180, Day 270, and Day 360 | 360 days
Proportion of participants with LDL-C greater than 80% of baseline value at Day 180, Day 210, Day 270, and Day 360 | 360 days
Duration of treatment for participants to return to 80% of baseline value or greater LDL-C or PCSK9 protein | 360 days
Proportion of participants who attained global lipid modification targets for level of ASCVD risk | 360 days
Number of participants with adverse events and injection site reactions, with abnormal vital signs, abnormal physical examination, abnormal 12-ECG, abnormal laboratory assessments | 360 days
ADA incidence | 360 days